CLINICAL TRIAL: NCT05134090
Title: Percutaneous Laparoscopy for Ovarian Tissue Cryopreservation: a Single-center Experience.
Brief Title: Percutaneous Laparoscopy for Ovarian Tissue Cryopreservation.
Status: Completed | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Benito Chiofalo, Principal Investigator, Regina Elena Cancer Institute
Other Study IDs: 1514/21
Record Dates: First submitted 2021-08-11; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Oncology; Fertility Issues; Surgery
Keywords: Percuvataneous laparoscopy; Ovarian Tissue Cryopreservation
MeSH Terms: conditions — Neoplasms; Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Percutaneous laparoscopy: Laparoscopy with percutaneous grasp (2.9 mm).
  Interventions: Device: Ovaian tissue explant
- Conventional laparoscopy: Conventional laparoscopy with conventional laparoscopic trocars (10 or 5 mm).
  Interventions: Device: Ovaian tissue explant

INTERVENTIONS:
Device: Ovaian tissue explant — Ovarian tissue explant for cryopreservation of ovarian tissue

SUMMARY:
To compare surgical outcomes of oncologic patients that underwent conventional laparoscopy and percutaneous laparoscopy for cryopreservation of ovarian tissue.

DETAILED DESCRIPTION:
This is a retrospective analysis to evaluate the efficacy and safety of percutaneous laparoscopy for the ovarian tissue explant in oncologic women. Surgical outcomes of patients that underwent percutaneous laparoscopy were compared with those of women that underwent conventional laparoscopy. Data from 2017 to 2021 were collected in a single Oncologic Center in Italy. The principal outcomes considered are post-operative pain, recovery time and aesthetic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Oncologic women with desire to preserve fertility

Exclusion Criteria:

* Ovarian explant with different techniques than laparoscopy

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with histological diagnosis of malignancy during reproductive age undergoing ovarian tissue explant for ovarian tissue cryopreservation, from Aug 2017 to Jun 2021.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | 0-1 and 2 days after surgery
  Post-operative pain is evaluated with VAS score ranging from 1 to 10 (higher score, maximum pain)
Aesthetic outcomes | minimum 3 months after surgery
  General satisfaction regarding aesthetic outcomes is collected with a satisfaction survey. The score ranged from 1 to 5, with 1 indicating "very dissatisfied" and 5 "very satisfied".

SECONDARY OUTCOMES:
Recovery time | Days
  Time from surgical intervention to discharge in days
Operative time | 1 day
  Time of operation in minutes
Blood loss | 1 day
  Entity of blood loss during surgery in ml
Surgical complications | 30 days
  The presence of absence of intra and post-operative complications (yes or not and type)

CONTACTS AND LOCATIONS:
Overall Officials: Benito Chiofalo, Principal Investigator — IRCCS "Regina Elena" National Cancer Institute
Locations (1):
- IRCCS "Regina Elena" National Cancer Institute, Rome, Lazio, Italy

REFERENCES:
- [Derived] Chiofalo B, Bruno V, Calandra M, Savone D, Mancini E, Baiocco E, Iacobelli M, Giannini A, Vizza E. Percutaneous-assisted laparoscopy for ovarian tissue cryopreservation: a single-center experience. Arch Gynecol Obstet. 2022 Oct;306(4):1329-1335. doi: 10.1007/s00404-022-06684-0. Epub 2022 Jul 10. PMID 35819490